CLINICAL TRIAL: NCT00004806
Title: Phase I Study of Liposome-Mediated Gene Transfer in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Purpose: Treatment
Other Study IDs: 199/11983; UAB-11983
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2011-03

CONDITIONS: Cystic Fibrosis
Keywords: cardiovascular and respiratory diseases; cystic fibrosis; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Diseases; Genetic Diseases, Inborn; Rare Diseases | interventions — Cystic Fibrosis Transmembrane Conductance Regulator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: Cystic fibrosis transmembrane conductance regulator

SUMMARY:
OBJECTIVES:

Evaluate the efficacy and safety of lipid-mediated transfer of the cystic fibrosis transmembrane conductance regulator gene to nasal epithelium in patients with cystic fibrosis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Cystic fibrosis transmembrane conductance regulator (CFTR) gene complexed with lipid is administered intranasally to the right inferior turbinate. Lipid without CFTR is administered to the left nostril as a control.

Cohorts of 3 patients are given successively lower doses of CFTR, each dose complexed with 500 micrograms of lipid.

Patients are followed at days 2-12, 15, and 21, then every 3-4 days for 3 weeks, every 2-3 weeks for 10 weeks, and every 3 months thereafter.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Cystic fibrosis (CF), i.e.: Sweat chloride greater than 60 mEq/L Clinical manifestations of CF Homozygous delta F508 mutation preferred Compound heterozygotes for F508 mutation with pancreatic insufficiency eligible FEV1 greater than 40% of predicted PO2 at least 60 mm Hg on room air No acute or recurrent sinusitis No obstructive nasal polyposis No pneumothorax or hemoptysis, e.g., more than 250 mL blood within 24-hour period, within past year No unstable lung disease with worsening pulmonary symptoms, arterial blood gas, or pulmonary function tests within 2 weeks prior to entry No pulmonary exacerbation within 4 weeks prior to entry --Prior/Concurrent Therapy-- At least 2 months since participation in any other clinical study At least 2 months since DNase At least 4 months since corticosteroids --Patient Characteristics-- Cardiac: No severe cardiac disease Other: No other severe organ system disease, e.g., juvenile-type diabetes mellitus No pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9
Dates: Start 1995-06; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J. Sorscher, Study Chair — University of Alabama at Birmingham